CLINICAL TRIAL: NCT01736683
Title: An Open-label, Randomized, Phase 2, Parallel, Dose-Ranging, Multicenter Study of Sotatercept for the Treatment of Patients With Anemia and Low or Intermediate-1 Risk Myelodysplastic Syndromes or Non-proliferative Chronic Myelomonocytic Leukemia (CMML)
Brief Title: Study of Sotatercept for the Treatment of Anemia in low-or Intermediate-1 Risk Myelodysplastic Syndromes (MDS) or Non-proliferative Chronic Myelomonocytic Leukemia (CMML)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7962-017; ACE-011-MDS-001 (Other: Celgene); 2012-002601-22 (EudraCT Number)
Record Dates: First submitted 2012-11-27; First posted 2012-11-29 (Estimated); Results first posted 2019-06-13 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Anemia; Myelodysplastic Syndromes; Chronic Myelomonocytic Leukemia; Low to Intermediate-1 MDS; Myelodysplastic Syndromes (MDS); Chronic Myelomonocytic Leukemia (CMML)
Keywords: ACE-011; anemia; dose-ranging; intermediate-1 risk myelodysplastic syndromes; low risk myelodysplastic syndromes (MDS); multicenter; open-label; parallel; phase 2; randomized; Sotatercept; Non-proliferative chronic myelomonocytic leukemia (CMML); hemoglobin; transfusions
MeSH Terms: conditions — Anemia; Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic | interventions — ACE-011

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Sotatercept 0.1 mg/kg (Experimental): Sotatercept 0.1 mg/kg
  Interventions: Drug: Sotatercept
- Sotatercept 0.3 mg/kg (Experimental): Sotatercept 0.3 mg/kg
  Interventions: Drug: Sotatercept
- Sotatercept 0.5 mg/kg (Experimental): Sotatercept 0.5 mg/kg
  Interventions: Drug: Sotatercept
- Sotatercept 1.0 mg/kg (Experimental): Sotatercept 1.0 mg/kg
  Interventions: Drug: Sotatercept
- Sotatercept 1.5 mg/kg (Experimental): Sotatercept 1.5 mg/kg
  Interventions: Drug: Sotatercept
- Sotatercept 2.0 mg/kg (Experimental): Sotatercept 2.0 mg/kg
  Interventions: Drug: Sotatercept

INTERVENTIONS:
Drug: Sotatercept — Sotatercept is supplied as a lyophilized powder that is reconstituted using Water for Injection (WFI) and administered as a subcutaneous injection (SC) injection by the study staff at the clinical site.
  Other Names: ACE-011; ActRIIA-IgG1Fc

SUMMARY:
The primary objective of this study is to determine a safe, tolerable and effective dose of sotatercept that results in the greatest frequency of improvement of anemia in patients diagnosed with low- or intermediate-1 risk myelodysplastic syndromes (MDS) or non-proliferative chronic myelomonocytic leukemia (CMML).

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18 years of age
* Documented diagnosis of myelodysplastic syndromes (MDS) or non-proliferative chronic myelomonocytic leukemia (CMML), white blood cells (WBC) ≤ 13,000 /mm^3, World Health Organization (WHO) that meets International Prognostic Scoring System (IPSS) criteria for low or intermediate-1 risk disease
* Anemia, Hemoglobin (Hgb) ≤ 9.0 g/dL or ≥ 2 units of Red Blood Cells (RBCs) within 84 days
* No response or loss of response to Erythropoiesis-Stimulating Agents (ESAs) or erythropoetin (EPO) > 500 mU/ml
* Eastern Cooperative Group (ECOG) score ≤2.
* Creatinine < 1.5 * Upper Limit of the Normal (ULN)
* Total bilirubin ≤3.0 mg/dL
* Aspartate aminotransferase (AST)/Serum glutamic oxaloacetic transaminase (SGOT) & Alanine Aminotransferase (ALT)/Serum Glutamic Pyruvic (SGPT) ≤3.0 * Upper Limit of Norma (ULN)
* Free of metastatic malignancy (other than MDS) for ≥2 years
* Highly effective methods of birth control for females and males

Exclusion Criteria:

* Chromosome 5q deletion
* Pregnant or breast feeding women and males who do not agree to use condom during the sexual contact with females of childbearing potential
* Major surgery within 30 days
* Incomplete recovery or incomplete healing of wounds from previous surgery
* Heart failure ≥3 (New York Heart Association (NYHA))
* Thromboembolic or myocardial infarction event within 6 months
* Concurrent anti-cancer cytotoxic chemotherapy
* History of severe allergic or anaphylactic reaction or hypersensitivity to recombinant protein
* Known positive for Human Immunovirus (HIV) or infectious Hepatitis type C or active infectious Hepatitis type B
* Clinically significant anemia unrelated to MDS
* Thrombocytopenia (<30,000/uL)
* Uncontrolled hypertension
* Treatment with another investigational drug or device within 28 days prior to Day 1
* Prior exposure to sotatercept (ACE-011)
* Any serious medical condition, lab abnormality or psychiatric illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2012-11-28 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Ito, MD, Study Director — Celgene Corporation
Locations (20):
- United States (13):
  - Rocky Mountain Cancer Center-Midtown, Denver, Colorado
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Johns Hopkins, Baltimore, Maryland
  - Dana-Farber / Harvard Cancer Institute, Boston, Massachusetts
  - Monter Cancer Center, North Shore LIJ Health Systems, Lake Success, New York
  - Columbia University Medical Center/New York-Presbyterian Hospital, New York, New York
  - The Cleveland Clinic Foundation Hematology and Medical Oncology Rm 35, Cleveland, Ohio
  - Sarah Cannon Research Inst, Nashville, Tennessee
  - Texas Oncology Round Rock Cancer Center - Round Rock, Round Rock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Texas Oncology, P.A. - Tyler, Tyler, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - Yakima Valley Memorial Hospital/ North Star Lodge, Yakima, Washington
- France (7):
  - Centre Hospitalier Universitaire d'Avicennes, Bobigny
  - Institute Paoli-Calmettes Service Haematology, BP 156,
  - CHRU de Lille-Hopital Claude Huriez Service des Maladies du Sang, Lille
  - CHRU Nantes, Nantes
  - Hopital Cochin Hematologie, Paris
  - Centre Henri Becquerel, Rouen
  - CHU Purpan, Toulouse

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Komrokji R, Garcia-Manero G, Ades L, Prebet T, Steensma DP, Jurcic JG, Sekeres MA, Berdeja J, Savona MR, Beyne-Rauzy O, Stamatoullas A, DeZern AE, Delaunay J, Borthakur G, Rifkin R, Boyd TE, Laadem A, Vo B, Zhang J, Puccio-Pick M, Attie KM, Fenaux P, List AF. Sotatercept with long-term extension for the treatment of anaemia in patients with lower-risk myelodysplastic syndromes: a phase 2, dose-ranging trial. Lancet Haematol. 2018 Feb;5(2):e63-e72. doi: 10.1016/S2352-3026(18)30002-4. Epub 2018 Jan 10. PMID 29331635

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were stratified by concentration of serum erythropoietin (EPO) (<500 versus ≥500 IU/L), by number of transfusions within 56 days of study enrollment (<4 versus ≥4 units of red blood cells) and assigned randomly to 0.1 mg/kg and 0.3 mg/kg arms.
Pre-assignment Details: Enrollment in the other arms (sotatercept 0.5, 1.0 and 2.0 mg/kg arms) commenced after the Steering Committee approved the higher doses based on the safety of preceding doses.
Groups:
- Sotatercept 0.1 mg/kg: Sotatercept 0.1 mg/kg administered via subcutaneous injection every third week (Q3W). Participants were randomized to either the 0.1 mg/kg arm or the 0.3 mg/kg arm. Efficacy and safety data were assessed by a Steering Committee. Based upon the occurrence of dose-limiting toxicity (DLT) in ≤ 1/5 subjects in Cycle 1 in the 0.1 mg/kg and 0.3 mg/kg treatment groups, the 0.5 mg/kg treatment group began inclusion in the randomization scheme.
- Sotatercept 0.3 mg/kg: Sotatercept 0.3 mg/kg administered via subcutaneous injection every third week (Q3W). Participants were randomized to either the 0.1 mg/kg arm or the 0.3 mg/kg arm. Efficacy and safety data were assessed by a Steering Committee. Based upon the occurrence of dose-limiting toxicity (DLT) in ≤ 1/5 subjects in Cycle 1 in the 0.1 mg/kg and 0.3 mg/kg treatment groups, the 0.5 mg/kg treatment group began inclusion in the randomization scheme.
- Sotatercept 0.5 mg/kg: Sotatercept 0.5 mg/kg administered via subcutaneous injection every third week (Q3W). Participants were randomized to one of the active treatment arms. Efficacy and safety data were assessed by a Steering Committee. Based upon the occurrence of dose-limiting toxicity (DLT) in ≤ 1/6 subjects in Cycle 1 in the 0.5 mg/kg treatment group, the 1.0 mg/kg treatment group began inclusion in the randomization scheme.
- Sotatercept 1.0 mg/kg: Sotatercept 1.0 mg/kg administered via subcutaneous injection every third week (Q3W). Participants were randomized to one of the active treatment arms. Efficacy and safety data were assessed by a Steering Committee. Based upon the occurrence of dose-limiting toxicity (DLT) in ≤ 1/6 subjects in Cycle 1 in the 1.0 mg/kg treatment group, the 2.0 mg/kg treatment group began inclusion in the randomization scheme. Following evaluation of all treatment group data by the Steering Committee, enrollment continued only in the 1.0 mg/kg arm because the arm had the greatest frequency of erythroid hematological improvement (HI-E).
- Sotatercept 2.0 mg/kg: Sotatercept 2.0 mg/kg administered via subcutaneous injection every third week (Q3W). Participants were randomized to one of the active treatment arms. Efficacy and safety data were assessed by a Steering Committee. The 2.0 mg/kg sotatercept dose was reduced to 1.5 mg/kg for ongoing and newly enrolled participants by protocol amendment.
Period: Overall Study
Arm/Group | Sotatercept 0.1 mg/kg | Sotatercept 0.3 mg/kg | Sotatercept 0.5 mg/kg | Sotatercept 1.0 mg/kg | Sotatercept 2.0 mg/kg
Started | 7 | 6 | 21 | 35 | 5
Completed | 0 (# who completed treatment) | 0 (# who completed treatment) | 0 (# who completed treatment) | 0 (# who completed treatment) | 0 (# who completed treatment)
Not Completed | 7 | 6 | 21 | 35 | 5
Not completed — Disease Relapse | 0 | 0 | 2 | 1 | 0
Not completed — Adverse Event | 0 | 2 | 2 | 3 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 3 | 1 | 1
Not completed — Lack of Therapeutic Effect | 7 | 4 | 13 | 20 | 1
Not completed — Progressive Disease | 0 | 0 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 1 | 9 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Sotatercept 0.1 mg/kg | Sotatercept 0.3 mg/kg | Sotatercept 0.5 mg/kg | Sotatercept 1.0 mg/kg | Sotatercept 2.0 mg/kg | Total
Number analyzed (Participants) | 7 | 6 | 21 | 35 | 5 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (8.3) | 75 (6.9) | 69 (8.0) | 71 (8.2) | 69 (13.0) | 70 (8.4)
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 3 | 0 | 7 | 6 | 1 | 17
  >=65 - <75 years | 2 | 3 | 8 | 17 | 2 | 32
  >=75 years | 2 | 3 | 6 | 12 | 2 | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 4 | 17 | 4 | 28
  Male | 4 | 6 | 17 | 18 | 1 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 0 | 0 | 2
  Not Hispanic or Latino | 7 | 6 | 13 | 19 | 4 | 49
  Unknown or Not Reported | 0 | 0 | 6 | 16 | 1 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 0 | 1
  White | 7 | 6 | 14 | 18 | 3 | 48
  More than one race | NA — not asked on CRF | NA — not asked on CRF | NA — not asked on CRF | NA — not asked on CRF | NA — not asked on CRF | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported | 0 | 0 | 7 | 16 | 1 | 24
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 6 | 15 | 18 | 4 | 50
  France | 0 | 0 | 6 | 17 | 1 | 24
Height [Mean (Standard Deviation); unit: meters] | 1.70 (0.110) | 1.75 (0.054) | 1.70 (0.093) | 1.68 (0.089) | 1.56 (0.043) | 1.68 (0.095)
Weight [Mean (Standard Deviation); unit: kg] | 85.3 (21.79) | 79.5 (13.90) | 77.9 (13.97) | 73.5 (15.55) | 56.4 (7.25) | 75.2 (16.14)
Erythropoietin level [Count of Participants; unit: Participants]
  <=200 mIU/mL | 2 | 3 | 6 | 16 | 2 | 29
  >200 to <=500 mIU/mL | 2 | 1 | 6 | 6 | 0 | 15
  >500 mIU/mL | 3 | 2 | 9 | 9 | 2 | 25
  Missing | 0 | 0 | 0 | 4 | 1 | 5
Red Blood Cell (RBC) Transfusion Burden Categories [Count of Participants; unit: Participants] — RBC units transfused during 56 days prior to the start of treatment.
  Participants
    < 4 units (Low Transfusion Burden) | 0 | 0 | 3 | 8 | 1 | 12
    >= 4 units (High Transfusion Burden) | 7 | 6 | 18 | 27 | 4 | 62
Number of Previous Erythropoiesis-Stimulating Agents (ESA) Therapies for Myelodysplastic Syndromes [Count of Participants; unit: Participants] — Myelodysplastic Syndromes (MDS)
  Participants
    0 ESA therapies | 1 | 0 | 1 | 0 | 0 | 2
    1 ESA therapy | 6 | 2 | 11 | 23 | 3 | 45
    2 ESA therapies | 0 | 4 | 8 | 10 | 2 | 24
    3 ESA therapies | 0 | 0 | 1 | 2 | 0 | 3
Number of Previous Non-ESA Agents for Myelodysplastic Syndromes (MDS) [Count of Participants; unit: Participants] — Erythropoiesis-Stimulating Agents (ESA)
  Participants
    0 non-ESA agents | 0 | 0 | 2 | 7 | 2 | 11
    1 non-ESA agent | 1 | 0 | 7 | 16 | 1 | 25
    2 non-ESA agents | 2 | 1 | 6 | 7 | 1 | 17
    3 non-ESA agents | 2 | 1 | 2 | 2 | 1 | 8
    4 non-ESA agents | 0 | 1 | 2 | 3 | 0 | 6
    5 non-ESA agents | 1 | 1 | 0 | 0 | 0 | 2
    >5 non-ESA agents | 1 | 2 | 2 | 0 | 0 | 5
International Prognostic Scoring System (IPSS) Risk Category [Count of Participants; unit: Participants] — The International Prognostic Scoring System for MDS (IPSS) assigns a prognostic score (0=good and increasing in risk by half-grades with the top score outlined below) for three prognostic variables: - Marrow blasts (score 0-2.0) - Karyotype (score 0-1.0) - Cytopenias: neutrophil, platelets, and Hg counts (score 0-0.5) The three individual scores are summed resulting in a full range of 0- 3.5 and placed into risk categories - 0 = low risk - 0.5-1.0 = intermediate-1 risk - 1.5-2.0 = intermediate-2 risk - >=2.5 = high risk
  Participants
    Low - 0 | 4 | 4 | 5 | 11 | 0 | 24
    Intermediate- 1: 0.5 to 1 | 3 | 2 | 16 | 24 | 5 | 50
    Intermediate- 2: 1.5 to 2 | 0 | 0 | 0 | 0 | 0 | 0
    High: >= 2.5 | 0 | 0 | 0 | 0 | 0 | 0
Erythropoietin Level [Count of Participants; unit: Participants]
  <=200 mIU/mL | 2 | 3 | 6 | 16 | 2 | 29
  >200 to <=500 mIU/mL | 2 | 1 | 6 | 6 | 0 | 15
  >500 mIU/mL | 3 | 2 | 9 | 9 | 2 | 25
  Missing | 0 | 0 | 0 | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Erythroid Hematological Improvement (HI-E) Starting Before the Completion of Five Cycles of Treatment (Responder Rate)
Description: The responder rate includes non-transfusion dependent efficacy (NTDE) participants and transfusion dependent efficacy (TDE) participants. For non-transfusion dependence efficacy (NTDE) participants who required < 4 units of RBCs in the 8 weeks prior to start of therapy, HI-E was defined as an increase of >=1.5 g/dL hemoglobin sustained for 56 days over a period of >=8 weeks. For transfusion dependence efficacy (TDE) participants who required >=4 units of RBCs in the 8 weeks prior to start of therapy, HI-E was defined as a decrease of >= 4 units of RBCs transfused sustained for 56 days over a period of 8 weeks.
Time Frame: Day 2 to Day 142
Population: Efficacy Evaluable Population: all participants who take at least one dose of study medication and have baseline and at least one post-baseline assessment of efficacy without major deviation from protocol.
Measure: Number; unit: percentage of participants
Arm/Group | Sotatercept 0.1 mg/kg | Sotatercept 0.3 mg/kg | Sotatercept 0.5 mg/kg | Sotatercept 1.0 mg/kg | Sotatercept 2.0 mg/kg
Number analyzed (Participants) | 7 | 6 | 21 | 35 | 5
percentage of participants
  All participants | 0 | 66.7 | 42.9 | 60.0 | 40.0
  NTDE subpopulation: number analyzed (Participants) | 0 | 0 | 3 | 8 | 1
  NTDE subpopulation |  |  | 33.3 | 62.5 | 100
  TDE subpopulation: number analyzed (Participants) | 7 | 6 | 18 | 27 | 4
  TDE subpopulation | 0 | 66.7 | 44.4 | 59.3 | 25.0

2. Secondary Outcome: Time to Erythroid Hematological Improvement (HI-E) Response
Description: Time to first response = start date of first response (HI-E) - first dose date + 1 day. For NTDE participants (who required < 4 units of RBCs in the 8 weeks prior to start of therapy), HI-E was defined as an increase of >=1.5 g/dL hemoglobin sustained for 56 days over a period of >=8 weeks. For TDE participants (who required >=4 units of RBCs in the 8 weeks prior to start of therapy), HI-E was defined as a decrease of >= 4 units of RBCs transfused sustained for 56 days over a period of 8 weeks.
Time Frame: Day 1 to Day 87
Population: Efficacy Evaluable Population of participants who responded
Measure: Median (Full Range); unit: days
Arm/Group | Sotatercept 0.1 mg/kg | Sotatercept 0.3 mg/kg | Sotatercept 0.5 mg/kg | Sotatercept 1.0 mg/kg | Sotatercept 2.0 mg/kg
Number analyzed (Participants) | 0 | 4 | 9 | 21 | 2
days
  All participants |  | 24.0 [2 to 44] | 1.0 [1 to 2] | 1.0 [1 to 86] | 48 [9 to 87]
  NTDE subpopulation: number analyzed (Participants) | 0 | 0 | 1 | 5 | 1
  NTDE subpopulation |  |  | 1.0 [1 to 1] | 1.0 [1 to 52] | 9.0 [9 to 9]
  TDE subpopulation: number analyzed (Participants) | 0 | 4 | 8 | 16 | 1
  TDE subpopulation |  | 24.0 [2 to 44] | 1.5 [1 to 2] | 1.5 [1 to 86] | 87 [87 to 87]

3. Secondary Outcome: Duration of Erythroid Hematological Improvement (HI-E)
Description: The duration of HI-E response for participants who responded was (the last date of the consecutive hemoglobin [Hgb] measurements of the first >=56 day interval) - (the first date of the consecutive Hgb measurements of the first >=56 day interval) + 1 day.
Time Frame: Day 1 to 183.7 weeks
Population: Efficacy Evaluable Population of participants who responded
Measure: Median (Full Range); unit: days
Arm/Group | Sotatercept 0.1 mg/kg | Sotatercept 0.3 mg/kg | Sotatercept 0.5 mg/kg | Sotatercept 1.0 mg/kg | Sotatercept 2.0 mg/kg
Number analyzed (Participants) | 0 | 4 | 9 | 21 | 2
days
  All participants |  | 62.5 [62 to 69] | 104.0 [56 to 1794] | 133.0 [58 to 1554] | 96.0 [58 to 134]
  NTDE subpopulation: number analyzed (Participants) | 0 | 0 | 1 | 6 | 1
  NTDE subpopulation |  |  | 79.0 [79 to 79] | 1043.0 [69 to 1554] | 134.0 [134 to 134]
  TDE subpopulation: number analyzed (Participants) | 0 | 4 | 8 | 16 | 1
  TDE subpopulation |  | 62.5 [62 to 69] | 105.5 [56 to 1794] | 96.5 [58 to 1033] | 58.0 [58 to 58]

4. Secondary Outcome: Time to Progression to Acute Myeloid Leukemia (AML) for Participants Who Had Progression
Description: Progression to AML used criteria by the International Working Group (IWG) Response Criteria in Myelodysplasia (Cheson, 2006). Progression is considered if any of the following are met: - >=50% increase in blasts - >=50% decrement from maximum remission/response levels in granulocytes or platelets - Reduction in Hgb concentration by >=2 g/dL - Transfusion dependence This outcome was defined as a Kaplan-Meier estimate however few participants progressed so a Kaplan-Meier analysis could not be performed. Disclosed are time to progression values only for participants who did progress to AML.
Time Frame: Day 1 to 183.7 weeks
Population: Efficacy Evaluable Population of participants who progressed to AML
Measure: Number; unit: weeks
Arm/Group | Sotatercept 0.1 mg/kg | Sotatercept 0.3 mg/kg | Sotatercept 0.5 mg/kg | Sotatercept 1.0 mg/kg | Sotatercept 2.0 mg/kg
Number analyzed (Participants) | 0 | 0 | 1 | 1 | 0
weeks |  |  | 45.6 | 78.0 |

5. Secondary Outcome: Time to Progression to Events of Higher Risk Myelodysplastic Syndromes (MDS) Using the International Prognostic Scoring System (IPSS) For Participants Who Had Progression
Description: Progression to events of higher risk MDS used criteria from the International Prognostic Scoring System for MDS (IPSS) which assigns a prognostic score (0=good and increasing in risk by half-grades with the top score outlined below) for three prognostic variables: - Marrow blasts (score 0-2.0) - Karyotype (score 0-1.0) - Cytopenias: neutrophil, platelets, and Hg counts (score 0-0.5) The three individual scores are summed resulting in a full range of 0- 3.5 and placed into risk categories 0 = low risk 0.5-1.0 = intermediate-1 risk 1.5-2.0 = intermediate-2 risk >=2.5 = high risk This outcome was defined as a Kaplan-Meier estimate however few participants progressed so a Kaplan-Meier analysis could not be performed. Data reported represent event times (weeks) for participants who did progress to higher risk MDS categories.
Time Frame: Day 1 to 257.3 weeks
Population: Efficacy Evaluable Population of participants who progressed to high risk MDS categories
Measure: Number; unit: weeks
Arm/Group | Sotatercept 0.1 mg/kg | Sotatercept 0.3 mg/kg | Sotatercept 0.5 mg/kg | Sotatercept 1.0 mg/kg | Sotatercept 2.0 mg/kg
Number analyzed (Participants) | 1 | 0 | 1 | 1 | 0
weeks | 15.1 |  | 24.7 | 67.4 |

6. Secondary Outcome: Kaplan-Meier Estimates for Progression-free Survival
Description: Participants who had disease progression were considered to have events. Participants who died without acute myeloid leukemia (AML) were also considered to have events with the event date as the date of death. Those who did not have disease progression and who were lost to follow-up were censored at the last known disease progression assessment date. Participants without disease progression at the last follow-up contact were censored at the date of the last follow-up contact date. Disease Progression to AML used criteria by the International Working Group (IWG) Response Criteria in Myelodysplasia (Cheson, 2006). Progression is considered if any of the following are met: - >=50% increase in blasts - >=50% decrement from maximum remission/response levels in granulocytes or platelets - Reduction in hemoglobin (Hgb) concentration by >=2 g/dL - Transfusion dependence
Time Frame: Day 1 to 257.3 weeks
Population: Efficacy Evaluable Population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Sotatercept 0.1 mg/kg | Sotatercept 0.3 mg/kg | Sotatercept 0.5 mg/kg | Sotatercept 1.0 mg/kg | Sotatercept 2.0 mg/kg
Number analyzed (Participants) | 7 | 6 | 21 | 35 | 5
weeks | 82.7 [15.1 to 82.7] | NA [91.1 to NA] — not enough events to allow for calculation | NA [58.6 to NA] — not enough events to allow for calculation | NA [NA to NA] — not enough events to allow for calculation | NA [79.9 to NA] — not enough events to allow for calculation

7. Secondary Outcome: Kaplan-Meier Estimates for Overall Survival (OS)
Description: OS was defined as the time between start of treatment and the death/censored date. Participants who died (regardless of the cause of death) were considered to have an event. Participants who were alive at the end of the study, and participants who were lost to follow-up, were censored at the last date when subjects were known to be alive.
Time Frame: Day 1 to 257.3 weeks
Population: Efficacy Evaluable Population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Sotatercept 0.1 mg/kg | Sotatercept 0.3 mg/kg | Sotatercept 0.5 mg/kg | Sotatercept 1.0 mg/kg | Sotatercept 2.0 mg/kg
Number analyzed (Participants) | 7 | 6 | 21 | 35 | 5
weeks | 82.7 [NA to NA] — not enough events to allow for calculation | NA [91.00 to NA] — not enough events to allow for calculation | NA [58.6 to NA] — not enough events to allow for calculation | NA [NA to NA] — not enough events to allow for calculation | NA [79.1 to NA] — not enough events to allow for calculation

8. Secondary Outcome: Pharmacokinetic Parameters of Sotatercept: Serum Concentration at Various Study Timepoints
Description: Maximum observed serum concentration, obtained directly from the observed concentration versus time data.
Time Frame: Cycle 1 Day 8 and !5 up to Cycle 2 Day 1
Population: Pharmacokinetic (PK) population includes participants with a sufficient amount of post-dose quantifiable PK sotatercept profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Sotatercept 0.5 mg/kg: Sotatercept 0.5 mg/kg administered via subcutaneous injection every third week (Q3W). Participants were randomized to one of the active treatment arms. Efficacy and safety data were assessed by a Steering Committee. Based upon the occurrence of dose-limiting toxicity (DLT) in ≤ 1/6 subjects in Cycle 1 in the 0.5 mg/ kg treatment group, the 1.0 mg/kg treatment group began inclusion in the randomization scheme.
- Sotatercept 1.0 mg/kg: Sotatercept 1.0 mg/kg administered via subcutaneous injection every third week (Q3W). Participants were randomized to one of the active treatment arms. Efficacy and safety data were assessed by a Steering Committee. Based upon the occurrence of dose-limiting toxicity (DLT) in ≤ 1/6 subjects in Cycle 1 in the 1.0 mg/ kg treatment group, the 2.0 mg/kg treatment group began inclusion in the randomization scheme. Following evaluation of all treatment group data by the Steering Committee, enrollment continued only in the 1.0 mg/kg arm because the arm had the greatest frequency of erythroid hematological improvement (HI-E).
Arm/Group | Sotatercept 0.1 mg/kg | Sotatercept 0.3 mg/kg | Sotatercept 0.5 mg/kg | Sotatercept 1.0 mg/kg | Sotatercept 2.0 mg/kg
Number analyzed (Participants) | 7 | 6 | 21 | 35 | 5
ng/mL
  Cycle 1 Day 8: number analyzed (Participants) | 7 | 6 | 21 | 34 | 5
  Cycle 1 Day 8 | 288.06 (70.94) | 1426.00 (27.76) | 2237.46 (40.77) | 6525.37 (28.31) | 12886.14 (30.47)
  Cycle 1 Day 15: number analyzed (Participants) | 6 | 6 | 21 | 33 | 5
  Cycle 1 Day 15 | 240.31 (75.32) | 1207.68 (16.14) | 1869.52 (36.97) | 5149.74 (36.04) | 8303.73 (43.57)
  Cycle 2 Day 1: number analyzed (Participants) | 6 | 6 | 20 | 35 | 5
  Cycle 2 Day 1 | 252.20 (28.43) | 957.58 (18.63) | 1323.91 (44.40) | 3467.58 (57.06) | 5329.63 (38.27)

9. Secondary Outcome: Participants With Treatment-Emergent Adverse Events (TEAE)
Description: An adverse event (AE) is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a subject during the course of a study. Treatment-emergent adverse events (TEAEs) are defined as any AE occurring or worsening on or after the first treatment of the study medication and within 42 days after the last dose. The severity of AEs was graded based on National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE), Version 4.0 and the scale: Grade 1 = Mild Grade 2 = Moderate Grade 3 = Severe Grade 4 = Life threatening Grade 5 = Death. Relation to study drug was determined by the investigator. A treatment-related TEAE is defined as TEAE which was considered to be related to the study drug and reported as 'Suspected' on the CRF. AEs with a missing relationship were treated as 'treatment-related' in data summaries.
Time Frame: Day 1 up to 59.2 months
Population: Safety population: all participants who receive at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Sotatercept 0.1 mg/kg | Sotatercept 0.3 mg/kg | Sotatercept 0.5 mg/kg | Sotatercept 1.0 mg/kg | Sotatercept 2.0 mg/kg
Number analyzed (Participants) | 7 | 6 | 21 | 35 | 5
Participants
  >= 1 Treatment-emergent adverse event (TEAE) | 6 | 4 | 20 | 34 | 5
  >=1 Treatment-related TEAE | 2 | 3 | 7 | 18 | 4
  >=1 Serious TEAE | 1 | 2 | 6 | 10 | 2
  >=1 Serious TEAE related to treatment | 0 | 0 | 0 | 0 | 1
  >=1 TEAE severity 3 or 4 | 1 | 2 | 9 | 13 | 2
  >=1 TEAE severity grade 3/4 related to treatment | 0 | 0 | 1 | 0 | 1
  >=1 TEAE leading to death | 0 | 1 | 0 | 0 | 0
  >=1 TEAE leading to dose reduction | 0 | 0 | 0 | 0 | 0
  >=1 TEAE leading to dose interruption | 0 | 1 | 2 | 9 | 1
  >=1 TEAE leading to dose interruption + reduction | 0 | 0 | 0 | 1 | 0
  >= 1 TEAE leading to drug discontinuation | 0 | 2 | 2 | 3 | 2

10. Secondary Outcome: Dose Limiting Toxicities (DLTs)
Description: The following were DLTs if the investigator suspected they were treatment related: 1. Increase to >= 140 mmHg systolic blood pressure 2. Increase to >=90 mmHg diastolic blood pressure 3. Increase to >=140 systolic and increase > 20 mmHg compared to baseline systolic 4. Increase to >=90 mmHg diastolic and increase > 20 mmHg compared to baseline diastolic 5. Introduction of new anti-hypertension medication during treatment 6. Increase in dose of baseline anti-hypertension medication during treatment 7. >= Grade 2 (moderate severity or worse) hypertension as an adverse event
Time Frame: Day 1 to 59.2 months
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Sotatercept 0.1 mg/kg | Sotatercept 0.3 mg/kg | Sotatercept 0.5 mg/kg | Sotatercept 1.0 mg/kg | Sotatercept 2.0 mg/kg
Number analyzed (Participants) | 7 | 6 | 21 | 35 | 5
Participants
  1. Increase to >= 140 mmHg systolic | 1 | 1 | 8 | 19 | 2
  2. Increase to >=90 mmHg diastolic | 0 | 0 | 2 | 2 | 1
  3. =140 systolic and increase > 20 mmHg base | 0 | 1 | 5 | 10 | 2
  4. >=90 mmHg diastolic and increase > 20 mmHg base | 0 | 0 | 2 | 2 | 1
  5. Introduction of new anti-hypertension med | 0 | 0 | 4 | 3 | 1
  6. Incre in dose of baseline anti-hypertension med | 0 | 0 | 0 | 0 | 0
  7.>= Grade 2 hypertension TEAE | 0 | 1 | 2 | 4 | 1

11. Secondary Outcome: Number of Participants Who Achieved Red Blood Cell (RBC)-Transfusion Independence During the Erythroid Hematological Improvement (HI-E) Interval
Description: Number of participants who achieved RBC-independence was defined as participants who required no RBC-transfusions during a 56-day interval of erythroid hematological improvement (HI-E). NTDE = non-transfusion dependence efficacy participants who required < 4 units of RBCs in the 8 weeks prior to start of therapy TDE = transfusion dependence efficacy participants who required >=4 units of RBCs in the 8 weeks prior to start of therapy
Time Frame: Day 2 to Day 142
Population: Efficacy Evaluable Population
Measure: Count of Participants; unit: Participants
Arm/Group | Sotatercept 0.1 mg/kg | Sotatercept 0.3 mg/kg | Sotatercept 0.5 mg/kg | Sotatercept 1.0 mg/kg | Sotatercept 2.0 mg/kg
Number analyzed (Participants) | 7 | 6 | 21 | 35 | 5
Participants
  All participants | 0 | 1 | 3 | 15 | 1
  NTDE subpopulation: number analyzed (Participants) | 0 | 0 | 3 | 8 | 1
  NTDE subpopulation |  |  | 1 | 6 | 1
  TDE subpopulation: number analyzed (Participants) | 7 | 6 | 18 | 27 | 4
  TDE subpopulation | 0 | 1 | 2 | 9 | 0

ADVERSE EVENTS:
Time Frame: Day 1 up to 60.7 months
Arm/Group | Sotatercept 0.1 mg/kg | Sotatercept 0.3 mg/kg | Sotatercept 0.5 mg/kg | Sotatercept 1.0 mg/kg | Sotatercept 2.0 mg/kg
All-Cause Mortality (participants affected / at risk) | 1/7 | 1/6 | 6/21 | 6/35 | 1/5
Serious Adverse Events (participants affected / at risk) | 1/7 | 2/6 | 6/21 | 10/35 | 2/5
Other Adverse Events (participants affected / at risk) | 6/7 | 4/6 | 18/21 | 32/35 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sotatercept 0.1 mg/kg (N=7) | Sotatercept 0.3 mg/kg (N=6) | Sotatercept 0.5 mg/kg (N=21) | Sotatercept 1.0 mg/kg (N=35) | Sotatercept 2.0 mg/kg (N=5)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Mass (General disorders) | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Escherichia pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Peritoneal abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 1
International normalised ratio increased (Investigations) | 0 | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Aortic stenosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sotatercept 0.1 mg/kg (N=7) | Sotatercept 0.3 mg/kg (N=6) | Sotatercept 0.5 mg/kg (N=21) | Sotatercept 1.0 mg/kg (N=35) | Sotatercept 2.0 mg/kg (N=5)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 2 | 1 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 2 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 2 | 0
Eye haemorrhage (Eye disorders) | 0 | 1 | 0 | 0 | 0
Eye inflammation (Eye disorders) | 0 | 0 | 0 | 0 | 1
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 2 | 0
Lacrimation increased (Eye disorders) | 0 | 1 | 2 | 0 | 0
Vitreous floaters (Eye disorders) | 1 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2 | 5 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 4 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 6 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 7 | 9 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 4 | 8 | 2
Salivary gland enlargement (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 3 | 9 | 1
Asthenia (General disorders) | 0 | 1 | 3 | 7 | 0
Chest discomfort (General disorders) | 1 | 0 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 3 | 0
Fatigue (General disorders) | 0 | 1 | 6 | 11 | 1
Gait disturbance (General disorders) | 0 | 1 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 1 | 0 | 3 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 2 | 0
Oedema (General disorders) | 0 | 0 | 0 | 1 | 1
Oedema peripheral (General disorders) | 2 | 2 | 6 | 11 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 1 | 4 | 1 | 1
Vessel puncture site swelling (General disorders) | 0 | 1 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 3 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 2 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 2 | 4 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 5 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 4 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 3 | 3 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 4 | 5 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 2 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 2 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 3 | 1
Creatinine renal clearance decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 2 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 2 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 4 | 8 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2 | 3 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 2 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Iron overload (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 4 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 4 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 3 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 4 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 2 | 1 | 6 | 2
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 3 | 0
Headache (Nervous system disorders) | 3 | 1 | 4 | 5 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 2 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 4 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 3 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 3 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0
Gynaecomastia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 6 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 6 | 2 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 3 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 8 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 4 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 3 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 2 | 4 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is > 1 year since study completion. Then, Investigator can publish if manuscript is submitted to Celgene 60 days prior to submission. If Celgene decides publication would hinder drug development, Investigator must delay submission for up to 90 additional days. Investigator must delete confidential information before submission and defer publication to permit patent applications.

DOCUMENTS (2):
  • Study Protocol (2015-08-04): https://cdn.clinicaltrials.gov/large-docs/83/NCT01736683/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-01): https://cdn.clinicaltrials.gov/large-docs/83/NCT01736683/SAP_001.pdf